CLINICAL TRIAL: NCT02322255
Title: A Natural History, Non-Interventional, Two-Part Study in Subjects With Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: A Natural History Study of Fibrodysplasia Ossificans Progressiva (FOP)
Status: Completed | Type: Observational
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Other Study IDs: PVO-1A-001
Record Dates: First submitted 2014-12-08; First posted 2014-12-23 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Natural History Study; Non-interventional Study; Observational Study; Heterotopic ossification; Fibrodysplasia Ossificans Progressiva; FOP disease progression; FOP flare-up progression; Clementia; Myositosis Ossificans Progressiva; Munchmeyer's Disease; FOP; Palovarotene
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples for biomarker and proteomic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Subjects: All subjects enrolled in the study.

SUMMARY:
Fibrodysplasia Ossificans Progressiva (FOP) is a rare, severely disabling disease characterized by painful, recurrent episodes of soft tissue swelling (flare-ups) that result in abnormal bone formation in muscles, tendons, and ligaments. Flare-ups begin early in life and may occur spontaneously or after soft tissue trauma, vaccinations, or influenza infections. Recurrent flare-ups progressively restrict movement by locking joints leading to cumulative loss of function and disability. This 3-year, non-interventional, two-part, natural history study is designed to gain insight into total body HO, FOP disease progression, the impact of FOP on subjects' physical functioning, and clinical features and biomarkers that may be useful in the diagnosis and monitoring of disease progression. This natural history study will also provide important information to inform the design of subsequent interventional trials.

DETAILED DESCRIPTION:
This is a multi-center, natural history, non-interventional, longitudinal study in subjects with classic FOP. A thorough baseline examination will be performed to determine the current status of disease in each subject. In Part A, two imaging modalities assessed total body HO at baseline, and the optimal method (low-dose whole body CT scan [excluding head]) will be employed in Part B for the balance of the study. Progression will be assessed at annual in-clinic visits (ie, at Months 12, 24, and 36) at which time the procedures conducted at the baseline visit will be repeated. In addition, site personnel will telephone subjects midway between the annual visits (ie, at Months 6, 18, and 30).

During the 36-month follow-up period, at least one new flare-up (with a maximum of one per year) will be carefully studied. An in-clinic visit will be performed within 14 days following the subject's identification of his/her flare-up. Additional visits at Day 42 and Day 84 (after the initial flare-up clinic visit) will be performed. An additional future visit may be scheduled after Day 84 at the discretion of the Principal Investigator (PI) for prolonged flare-ups. However, subjects with an eligible flare-up may elect to participate in an ongoing Clementia interventional study rather than continue in this natural history study.

ELIGIBILITY:
Inclusion Criteria:

- Subjects clinically diagnosed with classical FOP with documented R206H mutation or believed to carry the R206H mutation

Exclusion Criteria:

- Participation in an interventional clinical research study within the 4 weeks prior to enrollment

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with classic FOP (R206H mutation).
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total body burden of heterotopic ossification as assessed by the optimal imaging modality (low-dose whole body CT [excluding head]). | Month 36

SECONDARY OUTCOMES:
Change from baseline in physical function as assessed by range of motion. | Month 12, Month 24, and Month 36
Change from baseline in patient-reported use of assistive devices and adaptations. | Month 6, Month 12, Month 18, Month 24, Month 30, and Month 36
Change from baseline in a disease-specific patient-reported outcome measure (FOP-Physical Function Questionnaire [FOP-PFQ]). | Month 6, Month 12, Month 18, Month 24, Month 30, and Month 36
Change from baseline in a patient-reported measure of physical and mental health (PROMIS Global Health Scale). | Month 6, Month 12, Month 18, Month 24, Month 30, and Month 36
Change from baseline in biomarkers. | Month 12, Month 24, and Month 36
Flare-up progression as assessed by the change from baseline in heterotopic ossification at the flare-up site. | Flare-up initiation, Flare-up Days 42 and 84
Flare-up progression as assessed by the change from baseline in pain and swelling at the flare-up site. | Flare-up initiation, Flare-up Days 42 and 84
Flare-up progression as assessed by the change from baseline biomarkers. | Flare-up initiation, Flare-up Days 42 and 84
Flare-up progression as assessed by the change from baseline in physical function as assessed by range of motion. | Flare-up initiation, Flare-up Days 42 and 84
Flare-up progression as assessed by the change from baseline in a disease-specific patient-reported outcome measure (FOP-Physical Function Questionnaire [FOP-PFQ]). | Flare-up initiation, Flare-up Days 42 and 84
Flare-up progression as assessed by the change from baseline in a patient-reported outcome measure of physical and mental health (PROMIS Global Health Scale). | Flare-up initiation, Flare-up Days 42 and 84

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- United States (2):
  - University of California San Francisco, Division of Endocrinology and Metabolism, San Francisco, California
  - University of Pennsylvania, Center for FOP & Related Bone Disorders, Philadelphia, Pennsylvania
- Hospital Italiano de Buenos Aires, Department of Pediatrics, Buenos Aires, Argentina
- Queensland University of Technology (QUT) Institute of Health and Biomedical Innovation (IHBI), Woolloongabba, Queensland, Australia
- Hôpital Necker-Enfants Malades, Department of Genetics, Paris, France
- Gaslini Institute, Unit of Rare Diseases, Department of Pediatrics, Genoa, Italy
- The Royal National Orthopaedic Hospital, Brockley Hill, Stanmore, Middlesex, United Kingdom

REFERENCES:
- [Background] Connor JM, Evans DA. Fibrodysplasia ossificans progressiva. The clinical features and natural history of 34 patients. J Bone Joint Surg Br. 1982;64(1):76-83. doi: 10.1302/0301-620X.64B1.7068725.
- [Background] Zhang W, Zhang K, Song L, Pang J, Ma H, Shore EM, Kaplan FS, Wang P. The phenotype and genotype of fibrodysplasia ossificans progressiva in China: a report of 72 cases. Bone. 2013 Dec;57(2):386-91. doi: 10.1016/j.bone.2013.09.002. Epub 2013 Sep 17. PMID 24051199
- [Background] Cohen RB, Hahn GV, Tabas JA, Peeper J, Levitz CL, Sando A, Sando N, Zasloff M, Kaplan FS. The natural history of heterotopic ossification in patients who have fibrodysplasia ossificans progressiva. A study of forty-four patients. J Bone Joint Surg Am. 1993 Feb;75(2):215-9. doi: 10.2106/00004623-199302000-00008. PMID 8423182
- [Derived] Kaplan FS, Sponseller PD, Pignolo RJ. Thoracic Deformity in Fibrodysplasia Ossificans Progressiva. JBJS Rev. 2025 May 22;13(5). doi: 10.2106/JBJS.RVW.25.00042. eCollection 2025 May 1. PMID 40403126
- [Derived] Pignolo RJ, Al Mukaddam M, Baujat G, Brown MA, De Cunto C, Hsiao EC, Keen R, Le Quan Sang KH, Grogan DR, Marino R, Strahs AR, Kaplan FS. Study methodology and insights from the palovarotene clinical development program in fibrodysplasia ossificans progressiva. BMC Med Res Methodol. 2023 Nov 13;23(1):269. doi: 10.1186/s12874-023-02080-7. PMID 37957586
- [Derived] Pignolo RJ, Hsiao EC, Al Mukaddam M, Baujat G, Berglund SK, Brown MA, Cheung AM, De Cunto C, Delai P, Haga N, Kannu P, Keen R, Le Quan Sang KH, Mancilla EE, Marino R, Strahs A, Kaplan FS. Reduction of New Heterotopic Ossification (HO) in the Open-Label, Phase 3 MOVE Trial of Palovarotene for Fibrodysplasia Ossificans Progressiva (FOP). J Bone Miner Res. 2023 Mar;38(3):381-394. doi: 10.1002/jbmr.4762. Epub 2023 Jan 25. PMID 36583535
- [Derived] Pignolo RJ, Kimel M, Whalen J, Kawata AK, Artyomenko A, Kaplan FS. The Fibrodysplasia Ossificans Progressiva Physical Function Questionnaire (FOP-PFQ): A patient-reported, disease-specific measure. Bone. 2023 Mar;168:116642. doi: 10.1016/j.bone.2022.116642. Epub 2022 Dec 13. PMID 36526263
- [Derived] Warner SE, Kaplan FS, Pignolo RJ, Smith SE, Hsiao EC, De Cunto C, Di Rocco M, Harnett K, Grogan D, Genant HK. Whole-body Computed Tomography Versus Dual Energy X-ray Absorptiometry for Assessing Heterotopic Ossification in Fibrodysplasia Ossificans Progressiva. Calcif Tissue Int. 2021 Dec;109(6):615-625. doi: 10.1007/s00223-021-00877-6. Epub 2021 Jul 31. PMID 34331548
- [Derived] Kou S, De Cunto C, Baujat G, Wentworth KL, Grogan DR, Brown MA, Di Rocco M, Keen R, Al Mukaddam M, le Quan Sang KH, Masharani U, Kaplan FS, Pignolo RJ, Hsiao EC. Patients with ACVR1R206H mutations have an increased prevalence of cardiac conduction abnormalities on electrocardiogram in a natural history study of Fibrodysplasia Ossificans Progressiva. Orphanet J Rare Dis. 2020 Jul 29;15(1):193. doi: 10.1186/s13023-020-01465-x. PMID 32727600
- [Derived] Towler OW, Shore EM, Kaplan FS. Skeletal malformations and developmental arthropathy in individuals who have fibrodysplasia ossificans progressiva. Bone. 2020 Jan;130:115116. doi: 10.1016/j.bone.2019.115116. Epub 2019 Oct 23. PMID 31655222
- [Derived] Pignolo RJ, Baujat G, Brown MA, De Cunto C, Di Rocco M, Hsiao EC, Keen R, Al Mukaddam M, Sang KLQ, Wilson A, White B, Grogan DR, Kaplan FS. Natural history of fibrodysplasia ossificans progressiva: cross-sectional analysis of annotated baseline phenotypes. Orphanet J Rare Dis. 2019 May 3;14(1):98. doi: 10.1186/s13023-019-1068-7. PMID 31053156
- See also: website for the International FOP Association — http://www.ifopa.org